CLINICAL TRIAL: NCT04790214
Title: Effect of a Cardiac Rehabilitation Program on Chronic Heart Failure Patients in Yaoundé, Cameroon
Acronym: CARECA-CHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, CN NGANOU-GNINDJIO, MD, MSc, Dr, Principal investigator, Yaounde Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CARECA-CHF
Record Dates: First submitted 2021-02-25; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Chronic Heart Failure (CHF)
Keywords: Cardiac rehabilitation; Chronic Heart failure; Physical function; Cameroon

STUDY DESIGN:
Intervention Model Description: Patients with stable CHF in stage II or III of the New York Heart Association.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stable CHF patients (Experimental): Stable CHF patients on stage II/III based on the New York Heart Failure classification
  Interventions: Other: CHF Patients

INTERVENTIONS:
Other: CHF Patients — Cardiac rehabilitation program on CHF patients on 06-08 weeks. Program will include: physical aerobic re-training, therapeutic education on CHF, psychological follow-up, nutritional education

SUMMARY:
CARECA-CHF study is a non-randomized, prospective, single-arm study, enrolled ambulatory patients with stable chronic heart failure [New York Heart Association (NYHA) class II/III]. Patients will be followed-up during a period of 06-08 weeks. The aim of this study is to assess the effect of a cardiac rehabilitation program on patients with stable chronic heart failure in Yaoundé, Cameroon.

DETAILED DESCRIPTION:
CARECA-CHF study is a non-randomized, prospective, single-arm study, multicentric study. Patients with stable chronic heart failure [New York Heart Association (NYHA) class II/III] will be enrolled ambulatory. The program will take place during a period of 06-08 weeks.

The aim of this study is to assess the effect of a cardiac rehabilitation program on patients with stable chronic heart failure in a resource-limited country.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable chronic heart failure confirmed by a cardiac ultrasound and whose severity is rated stage II or III of NYHA followed at Yaoundé central hospital and Yaoundé general hospital;
* Stable under treatment;
* Whose cardiac ultrasound is less than six months old;
* Having given his free and informed consent.

Exclusion Criteria:

* Poor adherence to the cardiac rehabilitation program activities;
* Patients lost insight the program;
* Withdrawal of informed consent.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of VO2 max | 8 weeks
  Variation of VO2 max at baseline and the end of the study

SECONDARY OUTCOMES:
Variation in 6-minute walk test (6MWT) distance | 8 weeks
  Variation in 6MWT in meter distance from the baseline to week 6 or 8. By using pedometer
Variation of duration of exercise and maximum load | 8 weeks
  variation in duration of exercise and maximum load expressed by watt power
Variation in level of anxiety and depression; | 8 weeks
  Difference in level of anxiety and depression assessed by a questionnaire
Change in quality of life assessed by the Minnesota Living With Heart Failure Questionnaire (MLWHFQ) | 8 weeks
  Change in quality of life assessed by the Minnesota Living With Heart Failure Questionnaire (MLWHFQ) Minnesota Living With Heart Failure Questionnaire score at Week 8 adjusted for baseline
Variation of time-domain heart rate variability (HRV) parameters | 8 weeks
  Variation of time-domain heart rate variability parameters before and after the intervention
Variation of frequency-domain HRV parameters | 8 weeks
  variation of frequency-domain HRV parameters before and after the intervention. Variation of frequency-domain HRV parameters (HF, LF, LF/HF) before and after the intervention.
Variation of index hypopnea-apnea index | 8 weeks
  Variation of variation of index hypopnea-apnea after 6-8 weeks of aerobic training.
Variation of sleep quality index | 8 weeks
  variation of sleep quality index by Pittsburg questionnaire
Variation of nocturnal saturation | 8 weeks
  Variation of nocturnal saturation by oxymeter
Non adherence | 8weeks
  evaluation of non adherence by questionnaire at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Chris Nadège N Nganou-Gnindjio, MD, MAS, Principal Investigator — Yaounde Central Hospital
Locations (1):
- Dr Chris Nadège Nganou-Gnindjio, Yaoundé, Cameroon